CLINICAL TRIAL: NCT06635343
Title: The Effect of Inspiratory Muscle Training on Respiratory Function, Balance and Functional Capacity in Trainable Mentally Handicapped Children
Acronym: Inspiratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri University (Other)
Responsible Party: Principal Investigator, hanife abakay, Assoc Prof, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KayseriU
Record Dates: First submitted 2024-09-12; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Inspiratory Muscle Training
Keywords: Mental disability; breathing; inspiratory muscle training; balance
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPRP Group (Experimental): In the CPRP group, a chest physiotherapy program was given by the physiotherapist 5 days a week, for 8 weeks, including respiratory control, diaphragmatic breathing, thoracic expansion exercises, and physical activity recommendations, to be applied once a day.
  Interventions: Other: CPRP
- Experimental Inspiratuar Muscle Training Group (Experimental): The experimental group underwent inspiratory muscle training (IMT) with an inspiratory muscle training device 5 days a week for 8 weeks.
  Interventions: Other: Experimental Inspiratuar Muscle Training

INTERVENTIONS:
Other: CPRP — In the CPRP group, a chest physiotherapy program was given by the physiotherapist 5 days a week, for 8 weeks, including respiratory control, diaphragmatic breathing, thoracic expansion exercises, and physical activity recommendations, to be applied once a day.
  Arms: CPRP Group
Other: Experimental Inspiratuar Muscle Training — In the experimental group inspiratory muscle training was applied. Children in the experimental group started inspiratory muscle training at 30% of the measured intra-oral maximum inspiratory pressure (MIP) value with 30x2 breaths (1 minute rest between repetitions) for 5 days a week for 8 weeks. The training was carried out with MIP every week. The training was continued for a total of 8 weeks with 30% of the new value by re-measuring the MIP value every week The value was measured again and continued at 30% of the new value for a total of 8 weeks. During each inspiratory muscle training session, oxygen saturation data from the index finger were monitored with a pulse oximeter to prevent individuals from experiencing hypoxia
  Arms: Experimental Inspiratuar Muscle Training Group

SUMMARY:
Background: The aim of this study was to examine the effect of inspiratory muscle training on respiratory functions, balance and functional capacity in trainable mentally disabled individuals.

Methods: Within the scope of the study, 30 children, aged between 8 and 17 years, diagnosed with educable mental disabilities, were randomly divided into experimental and conventional physiotherapy rehabilitation program (CPRP) groups. Before and after the test, blood pressure, respiratory frequency, pulse oximetry heart rate and arterial oxygen saturation (SpO2) values, and Modified Borg scores for fatigue and dyspnea detection were recorded. Body composition analysis, respiratory function test, and 6-minute walk test (6MWT) were performed on all individuals. The experimental group underwent inspiratory muscle training (IMT) with an inspiratory muscle training device 5 days a week for 8 weeks. The CPRP group was given a chest physiotherapy program that included thoracic expansion exercises, postural drainage, cough improvement techniques and physical activity recommendations, to be applied once a day, 5 days a week, for 8 weeks. At the end of eight weeks, the evaluations were repeated. Data were analyzed using SPSS vn. 25.0 software. The Paired Samples t-test was used to determine within-group differences, and Two-way ANOVA was applied to repeated measures to compare time and group effects.

DETAILED DESCRIPTION:
This study was designed according to a controlled pre-test-post-test design. Voluntary consent forms were obtained from the subjects and their parents before the study. The study was conducted in accordance with the Declaration of Helsinki and the necessary Ethics Committee approval was received from XXXXX University Clinical Research Ethics Committee (Decision No: 2022\365). The total 30 individuals who met the inclusion criteria were allocated into two groups using a stratified block randomization procedure with opaque and sealed envelopes containing group allocation numbers obtained from a computer-generated random number table.The study included a total of 30 children aged 8-17 years with educable mental disabilities were randomly divided into experimental (n=15) and CPRP groups (n=15), who were educated at XXXXX Special Education Application Centre. The study inclusion criteria:

--defined as a primary diagnosis of educable mental retardation,

* age range between 8-17 years,
* not having a condition that prevents exercise,
* autism defined as educable mental retardation in children according to the diagnosis made by the Guidance and Research Centers, Down's syndrome, or epilepsy with seizures. There were no additional disabilities such as hearing impairment or orthopedic disability. Exclusion criteria:
* defined as mental retardation with a history of hospitalization within the last month.

Detailed medical histories, gender, age, weight, height and education level of all individuals were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion criteria were defined as a primary diagnosis of educable mental retardation,
* age range between 8-17 years,
* not having a condition that prevents exercise, autism defined as educable mental retardation in children according to the diagnosis made by the Guidance and Research Centers, Down's syndrome, or epilepsy with seizures.
* There were no additional disabilities such as hearing impairment or orthopedic disability.

Exclusion Criteria:

* mental retardation with a history of hospitalization within the last month.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
For the evaluation of functional capacity | 8 WEEKS
  The Six-Minute Walk Test (6MWT) was applied. Each subject was asked to walk as fast as possible at their own walking pace for 6 minutes in a 30-meter straight corridor. Before and after the test, blood pressure, respiratory frequency, pulse oximetry heart rate and arterial oxygen saturation (SpO2) values, and Modified Borg scores for fatigue and dyspnea detection were recorded. If there was a risky condition (excessive fatigue, too high pulse rate to continue walking, etc.) in the children, the test was terminated and the test was repeated when the child rested. At the end of the test, the 6MWT walking distance was recorded in meters. Of the two tests applied, the longer distance value for each individual was used for statistical analysis
To evaluate functional balance | 8 WEEKS
  the Pediatric Berg Balance Scale (PBBS) was applied, which is the version of the Berg Balance Scale (BBS) modified for children by Franjoine et al . The scale comprises 14 items including sitting balance, standing balance, sitting to standing/standing to sitting, transfers, stepping, reaching forward with outstretched arm, reaching the floor, turning, and placing foot on stool items. Each item ranked from 0 to 4. 0 shows inability to perform the instruction, while 4 shows the ability to perform without any difficulty. Maximum total score is 56. All evaluations were repeated at the end of 8 weeks for all the children in the experimental and CPRP groups.

SECONDARY OUTCOMES:
Respiratory muscle strength | 8 WEEKS
  Respiratory muscle strength evaluated by electronic intraoral pressure measuring device at the beginning and at the end of the 8-week training. (FVC, FEV1, TCL,, PEF, FEF, FEV1%)
Functional capacity | 8 WEEKS
  Functional capacity evaluated by 6-minute walking test at the beginning and at the end of the 8-week training.
Body Balance | 8 WEEKS
  body balance evaluated by paediatric berg balance test at the beginning and at the end of the 8-week training.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanife Abakay, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ulubay G, Kokturk N, Gorek Dilektasli A, Sen E, Ciftci F, Demir T, Yildiz O, Gemicioglu B, Saryal S. [Turkish Thoracic Society national spirometry and laboratory standards]. Tuberk Toraks. 2017 Jun;65(2):117-130. doi: 10.5578/tt.50748. Turkish. PMID 28990891
- See also: Ulubay G, Köktürk N, Görek Dilektaşlı A, et al. Turkish Thoracic Society national spirometry and laboratory standards. Turk Thorac J. 2017;65:117-30. — https://pubmed.ncbi.nlm.nih.gov/28990891/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28990891/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/28990891